CLINICAL TRIAL: NCT06620627
Title: Prospective Collection of Samples to Enable the Development of Natera Screening Assay for Early Cancer Detection (PROCEED-CRC)
Brief Title: Prospective Collection of Samples to Enable the Development of Natera Screening Assay for Early Cancer Detection
Acronym: PROCEED-CRC
Status: Recruiting | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 23-073-ECP
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer Screening
Keywords: colorectal cancer; colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants at average risk for colorectal cancer: Participants 40 years of age or older at time of consent, planning or intending to undergo asymptomatic screening colonoscopy.

SUMMARY:
The PROCEED-CRC study will prospectively collect blood samples from participants who are at average risk of colorectal cancer (CRC). Samples will be used for research use and the development of a blood-based CRC screening test.

DETAILED DESCRIPTION:
Participants who meet study inclusion criteria will be invited to enroll in the study and will provide written consent prior to study procedures. Participants will provide blood samples and will be required to have a colonoscopy performed within 120 days of their blood draw. No test results from the blood collection will be provided to participants or clinicians.

ELIGIBILITY:
Inclusion Criteria:

1. 40 years of age or older at time of consent.
2. Planning or intending to undergo asymptomatic screening colonoscopy.
3. Able to tolerate venipuncture for research draw(s).
4. Able and willing to provide blood samples within the 120 days prior to a colonoscopy procedure.
5. Willing and able to comply with the study visit schedule and study requirements.
6. Signed informed consent(s) must be obtained prior to participation in the study

Exclusion Criteria:

1. Any prior history of any kind of malignancy (exception: participants who have undergone surgical removal of skin squamous cell or basal cell cancer may be enrolled provided the procedure was completed at least 12 months prior to the date of provision of informed consent for the study)
2. Had a complete colonoscopy with adequate bowel preparation in the previous nine (9) years.
3. Undergoing diagnostic colonoscopy for investigation of symptoms such as unexplained and long-lasting diarrhea, overt rectal bleeding, e.g., hematochezia or melena, within the previous 30 days. (Blood on toilet paper, after wiping, does not constitute rectal bleeding)
4. Undergone colorectal cancer screening within the associated recommended intervals

   1. FOBT/FIT within the previous 12 months
   2. FIT-DNA test within the previous 36 months
   3. Blood-based CRC screening test within the previous 36 months
   4. Computed tomography colonography CTC within the previous 5 years
   5. Flexible sigmoidoscopy within the previous 5 years
5. Precancerous findings on most recent colonoscopy. This does not include benign, and/or hyperplastic polyps of any size (Note: Tissue biopsies that result in no histopathology findings are acceptable)
6. Had a prior colorectal resection for any reason other than sigmoid diverticular disease
7. Diagnosis or personal history of any of the following high-risk conditions for colorectal cancer:

   1. Inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohns disease
   2. Familial adenomatous polyposis (also referred to as FAP, including attenuated FAP)
   3. Hereditary non-polyposis colorectal cancer syndrome (also referred to as HNPCC or Lynch Syndrome)
   4. Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Gardners Syndrome, Turcots (or Crails) Syndrome, Cowdens Syndrome, Juvenile Polyposis, Cronkhite-Canada Syndrome, Neurofibromatosis and Familial Hyperplastic Polyposis

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 5,000 participants will enroll in the study in order to obtain 3,000 evaluable participants
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 12 months
  To collect samples for the research use and the development of a blood-based colorectal cancer screening test in the average risk population

CONTACTS AND LOCATIONS:
Locations (1):
- Natera, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No